CLINICAL TRIAL: NCT03377283
Title: Reduction of Ischemic-reperfusion Injury by Ex-vivo ATG-perfusion of Kidneys and Livers Prior Organ Transplantation
Brief Title: Peri-operative rATG-perfusion of Solid Transplants
Acronym: ATG-perfusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Katja Kotsch, Univ. Prof. Dr. Katja Kotsch, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UN4640
Record Dates: First submitted 2017-11-28; First posted 2017-12-19 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Organ Preservation Solutions
MeSH Terms: interventions — Antilymphocyte Serum; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AP-KTx/LTx (Active Comparator): Transplant recipients receiving an rATG-perfused kidney or liver
  Interventions: Biological: organ perfusion with rabbit anti-thymocyte globulin (rATG)
- CP-KTx/LTx (Placebo Comparator): Transplant recipients receiving a control-perfused kidney or liver.
  Interventions: Other: organ perfusion with saline

INTERVENTIONS:
Biological: organ perfusion with rabbit anti-thymocyte globulin (rATG)
  Arms: AP-KTx/LTx
Other: organ perfusion with saline
  Arms: CP-KTx/LTx

SUMMARY:
The increasing demand for organ transplantation and the shortage of available organs limit the success of organ transplantation programs. Consequently, acceptance of expanded criteria donor (ECD) organs with the consequences of higher risk of unfavorable transplantation outcome has become an increasing reality. Among the most prominent characteristics distinguishing ECD from Standard Criteria Donors (SCD) are risk factors including brain death (BD) or prolonged cold ischemia time (CI) amplifying ischemia reperfusion injury (IRI). Currently there are no standard regimens to improve the quality of ECD organs. Therefore, donor organ treatment might be a promising approach to substantially improve organ quality. It will be investigated whether the application of the peri-operative perfusion of kidneys and livers with the polyclonal antibody rabbit antithymocyte globulin (rATG) ameliorates IRI.

This trial is designed as a parallel armed randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving a kidney or liver transplant from deceased donors

Exclusion Criteria:

* Hepatitis C Virus/Human Immunodeficiency Virus, undergoing re-transplantation or under a public guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-08-17 (Actual); Primary Completion 2015-03-04 (Actual); Study Completion 2016-02-24 (Actual)

PRIMARY OUTCOMES:
Graft function | Day 7
  Graft function from baseline defined as serum creatinine (KTx arm) and aspartate transaminase (LTx arm).

SECONDARY OUTCOMES:
Graft function - creatinine | Days 1-7 post transplantation, month 3, month 6, month 12
  Graft function from baseline defined as serum creatinine (mg/dL) for the KTx arm.
Graft function - glomeralur filtration rate | Days 1-7 post transplantation, month 3, month 6, month 12
  Graft function from baseline defined as glomerular filtration rate (ml/min/1.73M2) for the KTx arm.
Graft function - serum urea | Days 1-7 post transplantation, month 3, month 6, month 12
  Graft function from baseline defined as serum urea (mg/dL) for the KTx arm.
Graft function - aspartate transaminase | Days 1-7 post transplantation, month 3, month 6, month 12
  Graft function from baseline defined as aspartate transaminase (mg/dL) for LTx arm.
Graft function - alanine transaminase | Days 1-7 post transplantation, month 3, month 6, month 12
  Graft function from baseline defined as alanine transaminase (mg/dL) for LTx arm.
Graft function - total serum bilirubin | Days 1-7 post transplantation, month 3, month 6, month 12
  Graft function from baseline defined as total serum bilirubin (mg/dL) for LTx arm.
Graft function - gamma-glutamyl transpeptidase | Days 1-7 post transplantation, month 3, month 6, month 12
  Graft function from baseline defined as gamma-glutamyl transpeptidase (mg/dL) for LTx arm.
Graft function - alkaline phosphatase | Days 1-7 post transplantation, month 3, month 6, month 12
  Graft function from baseline defined as alkaline phosphatase (mg/dL) for LTx arm.
Graft function - quick value | Days 1-7 post transplantation, month 3, month 6, month 12
  Graft function from baseline defined as quick value (%) for LTx arm.
Patient age - recipient | Day zero, at the time point of transplantation
  Recipient age (years).
Patient age - donor | Day zero, at the time point of transplantation
  Donor age (years).
BMI - recipient | Day zero, at the time point of transplantation
  Recipient BMI (weight (lb) / [height (in)]2 x 703).
BMI - donor | Day zero, at the time point of transplantation
  Donor BMI (weight (lb) / [height (in)]2 x 703).
Sex - recipient | Day zero, at the time point of transplantation
  Recipient sex.
Sex - donor | Day zero, at the time point of transplantation
  Donor sex.
Cold ischemia time | during transplantation
  Cold ischemia time (hours) from cross-clamping until start of anastomosis.
Warm ischemia time | during transplantation
  Warm ischemia time (hours) is the time from start of anastomosis until reperfusion.
Panel-reactive antibodies | Day zero, at the time point of transplantation
  Presence of panel-reactive antibodies (%) in KTx recipients.
Hospital stay | after transplantation
  Hospital stay (days) after transplantation
ICU stay | after transplantation
  Intensive care unit stay (days) after transplantation
Mortality | up to 12 month
  Death rate in the investigated groups.
Graft loss | up to 12 month
  Graft loss rate in the investigated groups.
HLA missmatch | Day zero, at the time point of transplantation
  Human leukocyte antigen mismatches in KTx recipients.
Delayed graft function | after transplantation
  Development of delayed graft function (requirement of dialysis within the first 7 post operative days) in KTx recipients.
Experimental analysis of perioperative taken biopsies | Peri-operatively (zero hour biopsy)
  mRNA Expression of pro-inflammatory and anti-inflammatory cytokine/chemokine pattern in biopsies will be analysed to evaluate immunactivation of the organ
Experimental analysis of peripheral blood monunuclear cells | prior transplantation, days 1-7 post transplantation, month 3, month 6, month 12 for lymphocyte expression analysis of peripheral blood
  Leukocyte-composition and activation pattern will be analysed from peripheral blood via flow cytometry of the recipient and the donor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ritschl PV, Gunther J, Hofhansel L, Kuhl AA, Sattler A, Ernst S, Friedersdorff F, Ebner S, Weiss S, Bosmuller C, Weissenbacher A, Oberhuber R, Cardini B, Ollinger R, Schneeberger S, Biebl M, Denecke C, Margreiter C, Resch T, Aigner F, Maglione M, Pratschke J, Kotsch K. Graft Pre-conditioning by Peri-Operative Perfusion of Kidney Allografts With Rabbit Anti-human T-lymphocyte Globulin Results in Improved Kidney Graft Function in the Early Post-transplantation Period-a Prospective, Randomized Placebo-Controlled Trial. Front Immunol. 2018 Aug 24;9:1911. doi: 10.3389/fimmu.2018.01911. eCollection 2018. PMID 30197644